CLINICAL TRIAL: NCT00264472
Title: A 2-Part Phase 1 Study Evaluating the Safety and Anti-Tumor Activity of ADH300004 (Eniluracil) Administered With 5-Fluorouracil (5-FU), and the Pharmacokinetics of 5-FU Given as: 5.0 mg ADH300004 With Escalating Doses of 5-FU Administered Orally 3 Weeks Out of 4 in Subjects With Refractory Solid Tumors (Part 1); or 5.0 mg ADH300004 With 5 FU Administered Orally as a Split Dose for 3 Weeks Out of 4 in Subjects With Hepatocellular Carcinoma, Non-Small Cell Lung Carcinoma, Gastric Cancer, Cervical Cancer, Prostate Cancer, or Breast Cancer (Part 2) (Adherex Protocol Number AHX-03-104)
Brief Title: A Study of 5 Fluorouracil and the Anti-Tumor Activity of ADH300004 and 5 Fluorouracil in Subjects With Incurable Solid Tumors
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of funds
Sponsor: Adherex Technologies, Inc. (Industry)
Responsible Party: Clinical Study Manager, Adherex Technoloogies
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Adherex Protocol # AHX-03-104
Record Dates: First submitted 2005-12-12; First posted 2005-12-13 (Estimated); Last update posted 2008-12-15 (Estimated); Status verified 2008-12

CONDITIONS: Neoplasms
Keywords: Cancer; Tumors; Neoplasms; Anticarcinogenic Agents; Antineoplastic Agents; Dihydrouracil Dehydrogenase (NADP)
MeSH Terms: conditions — Neoplasms | interventions — eniluracil

INTERVENTIONS:
Drug: ADH300004 — 5 mg

SUMMARY:
5 fluorouracil (5 FU), one of the most actively investigated anti-cancer drugs, is rapidly inactivated by the enzyme dihydropyrimidine dehydrogenase (DPD). ADH300004 blocks DPD. This study will test the safety and effects of oral ADH300004 14 hours prior to oral 5 FU in subjects with refractory solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* > or = 18 years of age
* Advanced or metastatic solid tumors:

Part 1: Histologically proven advanced or metastatic solid tumors refractory to standard therapy or for which no standard therapy exists

Part 2: Histologically proven advanced and/or metastatic solid tumor of one of the following 6 histologies, that is refractory to standard curative therapy or for which no curative therapy exists: HCC, NSCLC, gastric cancer, cervical cancer, prostate cancer, and breast cancer

* Radiologically documented measurable or evaluable (non-measurable) disease
* Adequate performance status and organ function, as evidenced by hematologic and biochemical blood testing
* Willing to not receive fluoropyrimidine containing chemotherapy for 8 weeks after the last dose of ADH300004 in this study

Exclusion Criteria:

* Cytotoxic chemotherapy, radiotherapy, or investigational drug within 28 days prior to study entry
* Non-cytotoxic cancer therapy within 14 days prior to study entry
* Portal hypertension with bleeding esophageal or gastric varices within the past 3 months
* Ascites that is refractory to conservative management
* Inability to take oral medication
* Active peptic ulcer disease
* Known hypersensitivity to 5-FU or ADH300004
* Stroke, major surgery, or other major tissue injury within 30 days before study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-01; Primary Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
Part 1: To determine the DLTs and MTD of the combination of ADH300004 and 5 FU administered orally in a weekly regimen, for 3 weeks with 1 week rest per cycle, in subjects with incurable solid tumors | 4 weeks
Part 2: To determine the DLTs and MTD of the combination of ADH300004 and 5-FU administered orally as a split dose for 3 out of 4 weeks in subjects with HCC, NSCLC, gastric cancer, cervical cancer, prostate cancer, and breast cancer | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Howard Burris, III, MD, Principal Investigator — SCRI Development Innovations, LLC
Locations (1):
- Sarah Cannon Research Institute, Nashville, Tennessee, United States

REFERENCES:
- See also: Adherex Technologies Inc. Corporate Homepage — http://www.adherex.com